CLINICAL TRIAL: NCT01095393
Title: National Data Bank for Rheumatic Disease (NDB) Registry Study of Safety in Rheumatoid Arthritis (RA) Patients Treated With Certolizumab Pegol (CZP; Cimzia®) and Non-biologic Disease-modifying Antirheumatic Drug (DMARD) Therapies
Brief Title: National Data Bank for Rheumatic Disease Registry Study of Safety in Patients With Rheumatoid Arthritis Treated With Cimzia® or Disease-modifying Antirheumatic Drugs (DMARDs)
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Collaborators: National Data Bank for Rheumatic Diseases (NDB) (Other)
Responsible Party: Sponsor
Other Study IDs: RA0005
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab Pegol; CZP; Cimzia®; NDB; registry
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Certolizumab pegol (CZP): Patients with RA receiving treatment with certolizumab pegol (CZP; Cimzia®)
- Non-biologic DMARD: Subjects with RA receiving treatment with non-biologic DMARD

SUMMARY:
Observational registry to assess the longer-term risk of serious infections and malignancies reported with TNFα-blocker therapy, as well as the longer-term risk of cardiovascular and thromboembolic events in adult Rheumatoid Arthritis (RA) patients treated with Cimzia® as compared to non-biologic DMARD-treated controls.

ELIGIBILITY:
Inclusion Criteria:

* RA and started treatment with certolizumab pegol (Cimzia®; CZP) or non-biologic DMARD within the last 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rheumatologist referral or patient direct enrollment
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with lymphoma | 6 years
  Number of participants with lymphoma during the observational period (up to 6 years)

SECONDARY OUTCOMES:
Number of participants with serious infections | 6 years
  Number of participants with serious infections during the observational period (up to 6 years)
Number of participants with non-lymphoma malignancies | 6 years
  Number of participants with non-lymphoma malignancies during the observational period (up to 6 years)
Number of participants with cardiovascular events | 6 years
  Number of participants with cardiovascular events during the observational period (up to 6 years)
Number of participants with thromboembolic events | 6 years
  Number of participants with thromboembolic events during the observational period (up to 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Wolfe, M.D., Study Director — National Data Bank for Rheumatic Disease